CLINICAL TRIAL: NCT01956162
Title: Evaluation of a New Customized Removable Device With Rocker Sole for Plantar Off-Loading "Orthèse Diabète" in the Healing of Foot Ulcers in Diabetic Patients
Brief Title: Evaluation of a New Device "Orthèse Diabète" in the Healing of Foot Ulcers in Diabetic Patients
Acronym: ORTHODIAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Proteor Group (Industry)
Collaborators: Société Francophone du Diabète (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROT-ORTHO-0913
Record Dates: First submitted 2013-09-26; First posted 2013-10-08 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Foot Ulcer, Diabetic
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group "Orthèse Diabète" (Experimental): Using "Orthèse Diabète", a new customized removable device with rocker sole for plantar off-loading
  Interventions: Device: Orthèse Diabète
- Control Group (Active Comparator): Using "Conventional devices", removable off-loading systems among the devices available in France
  Interventions: Device: "Conventional" Device

INTERVENTIONS:
Device: Orthèse Diabète — The device ensures the discharge of the wound by the excavation of the orthopedic insole facing the wound and the load distribution in the healthy areas.
  Arms: Group "Orthèse Diabète"
Device: "Conventional" Device — Standard (e.g.: CHUT, BAROUK, Tera-Diab, Sanital, Teraheel, Aircast boots, Walker Stabil D, etc.), or customized (orthopedic insole, Ransart boot, D.T.A.C.P., etc.) removable off-loading systems
  Arms: Control Group

SUMMARY:
Multi-center trial, randomized in 2 parallel groups, open label, with a blinded adjudication committee (PROBE methodology), comparing "Orthèse Diabète" with "conventional" removable devices in terms of healing of ulcers.

- Primary objective: Evaluate the efficiency of "Orthèse Diabète" compared to "conventional" removable devices, in terms of the proportion of diabetic patients whose principal ulcer will heal completely at 3 months.

DETAILED DESCRIPTION:
1. Secondary objectives

   1. Proportion of patients whose principal ulcer will heal completely at 1, 2 and 6 months
   2. Proportion of patients in whom all initial plantar ulcers will heal completely at 1, 2, 3 and 6 months
   3. Percentage of area decrease of the plantar ulcers at 1, 2, 3 and 6 months
   4. Time to healing of the principal ulcer
   5. Appearance of new ulcers
   6. Requirement for amputation
   7. Incidence of the infectious complications
   8. Adherence of wearing
   9. Patient's satisfaction with the prescribed device
2. Population

   1. 13 centers/116 patients monitored for a period of 6 months maximum
   2. Experimental Group: "Orthèse Diabète" a plantar off-loading custom-made removable device
   3. Control group: "Conventional" removable off-loading systems among the devices available in France.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetic patients diagnosed according to the ADA experts consensus [ADA 1997]
* Over 18 years of age
* With a sensory neuropathy (abnormal 10 g monofilament test, i.e. not perceived at least 2 times in 1 of the 3 areas explored : pulp of the great toe, 1st and 5th metatarsal heads)
* Without a severe arteriopathy defined by : ABI < 0,7 and/or TcPO2 < 30 mm Hg and/or big toe pressure < 30 mm Hg
* with one or more plantar ulcerations with an area > 0,25 cm² or an amputation (toes or transmetatarsal) open or sutured
* not requiring a contralateral off-loading device
* Informed about the study and having given their informed and written consent to participate
* registered with a social security scheme or with the CMU (beneficiary or entitled recipient)
* having undergone a medical exam
* not included in another protocol throughout the study

Exclusion Criteria:

* Severe skin or osteoarticular infection requiring a parenteral antibiotic therapy or surgery
* Large ulcer of the ipsilateral leg > 20 cm2 of area
* Contralateral above heel amputation
* Intercurrent disease prohibiting participation in the protocol
* Weight over 130 Kg
* Person under tutorship or under curatorship
* Loss of functional and/or neuropsychological autonomy
* Pregnant or likely to be pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2013-10; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficiency of "Orthèse Diabète" compared to "conventional" removable devices, in terms of the proportion of diabetic patients whose principal ulcer will heal completely. | At 3 months
  Evaluated by taking photographs, measuring the ulcer area (using Digital Photo Planimetry DPP and the software Tracer.exe). Full healing defined by the adjudication committee based on the analysis of the photographs.

SECONDARY OUTCOMES:
Proportion of patients whose principal plantar ulcer will be fully healed | At 1, 2 and 6 months
  Evaluated by taking photographs, measuring the ulcer area (using Digital Photo Planimetry DPP and the software Tracer.exe). Full healing defined by the adjudication committee based on the analysis of the photographs.
Proportion of patients whose all initial plantar ulcers will be fully healed. | At 1, 2, 3 and 6 months
  Evaluated by taking photographs, measuring the ulcer area (using Digital Photo Planimetry DPP and the software Tracer.exe). Full healing defined by the adjudication committee based on the analysis of the photographs.
Percentage decrease of the ulcer area | At 1, 2, 3 and 6 months
  The area is evaluated by the last measurement undertaken during the trial or prior to a serious event (death, amputation, orthopedic or vascular surgery).
Time to healing of the principal ulcer | From the patient's off-loading device delivery visit to the date of healing validated by the adjudication committee
Appearance of new ulcers on the affected foot and/or contralateral | 6 months
  The following elements will be specified: cause, side, location, severity, treatment used
Requirement for amputation | 6 months
  The following elements will be specified: date, side and level.
Incidence of infectious complications | 6 months
  This covers cutaneous infections (abscess and lymphangitis, erysipelas, hypodermitis, necrotizing fasciitis, gas gangrene), bone infections (osteitis, arthritis, osteoarthritis) or systemic infections requiring antibiotic therapy (oral or parenteral) or surgery.
Observance of the equipment | 6 months
  Daily wear will be evaluated in the 2 groups through a semi-quantitative questionnaire provided to the patient at every visit. This evaluation will be supplemented with readings of the thermal sensor in the "Orthèse Diabète " group
Patients satisfaction with the prescribed device | At 3 months
  Evaluated with the "QUEST ESAT" questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kamel Mohammedi, Diabetology, Principal Investigator — Bichat Hospital
Locations (1):
- Bichat Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Malgrange D. [Physiopathology of the diabetic foot]. Rev Med Interne. 2008 Sep;29 Suppl 2:S231-7. doi: 10.1016/S0248-8663(08)73950-X. French. PMID 18822248
- [Background] Cavanagh PR, Lipsky BA, Bradbury AW, Botek G. Treatment for diabetic foot ulcers. Lancet. 2005 Nov 12;366(9498):1725-35. doi: 10.1016/S0140-6736(05)67699-4. PMID 16291067
- [Background] Ramsey SD, Newton K, Blough D, McCulloch DK, Sandhu N, Reiber GE, Wagner EH. Incidence, outcomes, and cost of foot ulcers in patients with diabetes. Diabetes Care. 1999 Mar;22(3):382-7. doi: 10.2337/diacare.22.3.382. PMID 10097914
- [Background] Muller IS, de Grauw WJ, van Gerwen WH, Bartelink ML, van Den Hoogen HJ, Rutten GE. Foot ulceration and lower limb amputation in type 2 diabetic patients in dutch primary health care. Diabetes Care. 2002 Mar;25(3):570-4. doi: 10.2337/diacare.25.3.570. PMID 11874949
- [Background] Detournay B, Cros S, Charbonnel B, Grimaldi A, Liard F, Cogneau J, Fagnani F, Eschwege E. Managing type 2 diabetes in France: the ECODIA survey. Diabetes Metab. 2000 Nov;26(5):363-9. PMID 11119015
- [Background] Detournay B, Raccah D, Cadilhac M, Eschwege E. Epidemiology and costs of diabetes treated with insulin in France. Diabetes Metab. 2005 Jun;31(3 Pt 2):3-18. PMID 16142041
- [Background] Malgrange D, Richard JL, Leymarie F; French Working Group On The Diabetic Foot. Screening diabetic patients at risk for foot ulceration. A multi-centre hospital-based study in France. Diabetes Metab. 2003 Jun;29(3):261-8. doi: 10.1016/s1262-3636(07)70035-6. PMID 12909814
- [Background] Apelqvist J, Larsson J, Agardh CD. Long-term prognosis for diabetic patients with foot ulcers. J Intern Med. 1993 Jun;233(6):485-91. doi: 10.1111/j.1365-2796.1993.tb01003.x. PMID 8501419
- [Background] Boulton AJ, Vileikyte L, Ragnarson-Tennvall G, Apelqvist J. The global burden of diabetic foot disease. Lancet. 2005 Nov 12;366(9498):1719-24. doi: 10.1016/S0140-6736(05)67698-2. PMID 16291066
- [Background] Moxey PW, Hofman D, Hinchliffe RJ, Jones K, Thompson MM, Holt PJ. Epidemiological study of lower limb amputation in England between 2003 and 2008. Br J Surg. 2010 Sep;97(9):1348-53. doi: 10.1002/bjs.7092. PMID 20632310
- [Background] Resnick HE, Carter EA, Sosenko JM, Henly SJ, Fabsitz RR, Ness FK, Welty TK, Lee ET, Howard BV; Strong Heart Study. Incidence of lower-extremity amputation in American Indians: the Strong Heart Study. Diabetes Care. 2004 Aug;27(8):1885-91. doi: 10.2337/diacare.27.8.1885. PMID 15277412
- [Background] Fosse S, Hartemann-Heurtier A, Jacqueminet S, Ha Van G, Grimaldi A, Fagot-Campagna A. Incidence and characteristics of lower limb amputations in people with diabetes. Diabet Med. 2009 Apr;26(4):391-6. doi: 10.1111/j.1464-5491.2009.02698.x. PMID 19388969
- [Derived] Potier L, Francois M, Dardari D, Feron M, Belhatem N, Nobecourt-Dupuy E, Dolz M, Bordier L, Ducloux R, Chibani A, Eveno DF, Crea Avila T, Sultan A, Baillet-Blanco L, Rigalleau V, Gand E, Saulnier PJ, Velho G, Roussel R, Pellenc Q, Dupre JC, Malgrange D, Marre M, Mohammedi K; ORTHODIAB study group. Comparison of a new versus standard removable offloading device in patients with neuropathic diabetic foot ulcers: a French national, multicentre, open-label randomized, controlled trial. BMJ Open Diabetes Res Care. 2020 May;8(1):e000954. doi: 10.1136/bmjdrc-2019-000954. PMID 32393479
- [Derived] Mohammedi K, Potier L, Francois M, Dardari D, Feron M, Nobecourt-Dupuy E, Dolz M, Ducloux R, Chibani A, Eveno DF, Crea Avila T, Sultan A, Baillet-Blanco L, Rigalleau V, Velho G, Tubach F, Roussel R, Dupre JC, Malgrange D, Marre M. The evaluation of off-loading using a new removable oRTHOsis in DIABetic foot (ORTHODIAB) randomized controlled trial: study design and rational. J Foot Ankle Res. 2016 Aug 22;9(1):34. doi: 10.1186/s13047-016-0163-4. eCollection 2016. PMID 27555884